CLINICAL TRIAL: NCT03382015
Title: Randomized, Double-Blind, Placebo-Controlled, Two-Period Crossover Study to Evaluate the Effect of BKR-013 on Average Daily Glucose Levels in Type 2 Diabetes Patients
Brief Title: Effect of BKR-013 on Average Daily Glucose Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioKier Inc. (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: CL-201; 4R44DK107080-02 (NIH)
Record Dates: First submitted 2017-12-11; First posted 2017-12-22 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Receives 28 days of active test product (BKR-013) in Part 1 of the study and receives 28 days of placebo in Part 2 of the study, following a washout period.
  Interventions: Other: BKR-013 or Placebo
- Group 2 (Placebo Comparator): Receives 28 days of placebo in Part 1 of the study and receives 28 days of active test product (BKR-013) in Part 2 of the study, following a washout period.
  Interventions: Other: BKR-013 or Placebo

INTERVENTIONS:
Other: BKR-013 or Placebo — Encapsulated L-glutamine

SUMMARY:
The purpose of this study is to evaluate the effect of BKR-013 on average daily glucose (ADG) levels in type 2 diabetes (T2D) subjects during 28 days of either placebo or active test product administration. Subjects will serve as their own controls in this crossover design, and ADG will be compared while a subject is on active test product versus while they received placebo test product.

DETAILED DESCRIPTION:
The study consists of a screening period followed by a 28-day treatment period, a 3 to 5 week washout period, and a second treatment period. All subjects receive both active test product and placebo, but the order in which they receive them (Part 1 or Part 2 of the study) is randomized in this single crossover study. Fourteen subjects will be randomized to ensure that 10 subjects complete both Part 1 and Part 2 of the study.

There are a total of 7 study visits including screening. In Part 1, Visits 2, 3 and 4 occur 2 weeks apart; in Part 2, Visits 5, 6 and 7 also occur 2 weeks apart. Visits 4 and 7 are overnight visits during which time hunger and satiety will be assessed and a Mixed Meal Tolerance Test (MMTT) will be performed after an overnight fast. The MMTT requires use of an indwelling IV catheter so that 11 blood draws can be more comfortably obtained over a period of 4 hours.

Subjects will be required to wear a glucose monitoring sensor during Part 1 and Part 2 of the study in order to obtain ADG levels.

Routine chemistry and hematology tests are done at 4 timepoints during the study. An ECG and physical exam is performed at screening.

A rapid HbA1c will only be tested at screening; if the value is between 6.5% and 10.5%, all other screening procedures will be performed; if the HbA1c value is not within the qualifying range, the subject will be considered a screen failure and no other screening procedures will be performed.

Subjects are required to keep a daily diary to document dosing (twice daily), medication changes and any adverse events.

Safety tests include chemistry/hematology, vital signs and adverse events.

Subjects with type 2 diabetes must be under the care of a healthcare professional to take part in this study. The test product BKR-013 is not designed to treat diabetes; it is being evaluated as a non-prescription medical food for nutritional use in managing glucose levels.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 18 and 70 years at the time of screening, inclusive
2. Diagnosed with T2D and under the care of a healthcare professional for its management
3. HbA1c 6.5-10.5%, inclusive
4. Has given written informed consent to participate in this study
5. Agrees to comply with all study requirements, including maintaining current diet and exercise routine and current prescription medications for the duration of the study
6. Willing to wear a Continuous Glucose Monitoring (CGM) sensor continuously for 28 days during each of the two test periods
7. Willing to complete two 28-day test periods (separated by a wash-out period of 21 to 35 days) and participate in the study for a total duration of up to 18 weeks.

Exclusion Criteria:

1. Type 1 diabetes
2. History of bariatric or intestinal surgery
3. Active gastrointestinal disease including but not limited to irritable bowel syndrome, inflammatory bowel disease (e.g., Crohn's disease and ulcerative colitis), diverticulitis, gastroparesis, or chronic/frequent diarrhea or chronic/frequent constipation
4. Active and clinically significant hepatic, pancreatic disease, or renal disease as determined by the investigator
5. History of significant heart disease, including congestive heart failure, prior MI, chronic atrial or ventricular fibrillation, coronary artery disease, cerebral vascular disease or other cardiovascular disease, that in the opinion of the investigator should exclude the subject from the study
6. Severely uncontrolled hypertension at screening defined as a systolic blood pressure > 180 mmHg or a diastolic blood pressure > 110 mmHg on the average of two seated measurements after being at rest for at least 5 minutes
7. Uncontrolled hyperthyroidism or hypothyroidism, or other significant thyroid disease
8. Active significant infection as determined by the investigator
9. Known allergy to L-glutamine or any of the components of the capsules
10. Participation in a clinical trial and/or treatment with an investigational drug during the 30 days before screening, or within 5 half-lives of receipt of an investigational drug or twice the duration of the biological effect of any investigational drug (whichever is longer)
11. Allergy or intolerance to Boost® High Protein drink
12. Magnetic Resonance Imaging (MRI), Computed Tomography (CT) scan or high-frequency electrical heat (diathermy) treatment scheduled during either of the 4-week test periods that a subject is wearing CGM sensor.
13. Pregnant, nursing, or trying to become pregnant
14. Presence of pitting edema on physical exam
15. High fiber diet
16. In the investigator's judgment, the subject is not suitable for the study for any other reason or cannot commit to the requirements of the study.
17. Subject is taking one or more of the excluded therapies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Average Daily Glucose Levels | After 28 days of treatment in Part 1 and in Part 2
  Intra-patient comparison of ADG in Part 1 vs Part 2

SECONDARY OUTCOMES:
Glucose >180 mg/dL | After 28 days of treatment in Part 1 and in Part 2
  Percent of each 24-hour period that a subject's glucose is >180 mg/dL
Triglycerides | After 28 days of treatment in Part 1 and in Part 2
  Differences in fasting triglycerides between active test product and placebo

CONTACTS AND LOCATIONS:
Overall Officials: George R Szewczyk, PhD, Study Director — BioKier Inc.
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No